CLINICAL TRIAL: NCT00989950
Title: Open Label Study of the Effect of Individualizing Daytrana Wear-times on Sleep in Children 6-12 Years Old With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Study of the Effect of Individualizing Daytrana Wear-times on Sleep in Children With ADHD
Acronym: Daytsleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cox Health Systems (Other)
Responsible Party: Principal Investigator, Arie Ashkenasi, MD, Staff Neurologist, Cox Health Systems
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: cox002; shire IND#54,732 (Other: Shire Pharmaceuticals)
Record Dates: First submitted 2009-09-30; First posted 2009-10-06 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; INSOMNIA
Keywords: daytrana; sleep latency; adhd rating scales; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Daytrana 9 hr wear (Experimental)
  Interventions: Drug: Daytrana
- Daytrana 10 hr wear (Experimental)
  Interventions: Drug: Daytrana
- Daytrana 11 hr wear (Experimental)
  Interventions: Drug: Daytrana
- Daytrana 12 hr wear (Experimental)
  Interventions: Drug: Daytrana

INTERVENTIONS:
Drug: Daytrana — Daytrana patch 10-30 mg administered once daily for 9hr
  Other Names: methylphenidate transdermal system
  Arms: Daytrana 9 hr wear
Drug: Daytrana — Daytrana 10-30 mg worn once daily for 10 hr wear
  Other Names: methylphenidate transdermal system
  Arms: Daytrana 10 hr wear
Drug: Daytrana — Daytrana 10-30 mg worn once daily for 11 hr
  Other Names: methylphenidate transdermal system
  Arms: Daytrana 11 hr wear
Drug: Daytrana — Daytrana 10-30 mg worn once daily for 12 hrs
  Arms: Daytrana 12 hr wear

SUMMARY:
Methylphenidate may improve sleep in children with ADHD. By leaving Daytrana (methylphenidate) patch for a longer time then 9 hours, many children report short sleep latencies and better quality of sleep.

DETAILED DESCRIPTION:
Once the optimal dose of Daytrana that controlled the ADHD symptoms is established. The patch will be removed 1, 2, and 3 hours before bed time in a random fashion, at weekly intervals, and parents will keep a sleep diary.

25 patients will be enrolled in order to obtain statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* ADHD without significant comorbidity

Exclusion Criteria:

* Cardiac disorder
* Hypertension
* Thyroid disease
* Glaucoma
* History of sudden death, motor tics and/or Tourette's syndrome
* Hypersensitivity to methylphenidate

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: arie ashkenasi, Principal Investigator — pediatric neurology of the ozarks
Locations (1):
- Pediatric Neurology of the Ozarks, Springfield, Missouri, United States

REFERENCES:
- [Result] Ashkenasi A. Effect of transdermal methylphenidate wear times on sleep in children with attention deficit hyperactivity disorder. Pediatr Neurol. 2011 Dec;45(6):381-6. doi: 10.1016/j.pediatrneurol.2011.09.003. PMID 22115000

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Sequence 1: Daytrana 10-30 mg worn 10 hrs, 12 hrs, 9 hrs then 11 hrs daily each period lasting Monday-Thursday of each week, followed by 12 hr daily wear on Fri-Sun
- Group Sequence 2: Daytrana 10-30 mg worn 11 hrs, 9 hrs, 12 hrs then 10 hrs daily each period lasting Monday-Thursday of each week, followed by 12 hr daily wear on Fri-Sun
- Group Sequence 3: Daytrana 10-30 mg worn 9 hrs, 10 hrs, 11 hrs, then 12 hrs daily each period lasting Monday-Thursday of each week, followed by 12 hr daily wear on Fri-Sun
- Group Sequence 4: Daytrana 10-30 mg worn 12 hrs, 11 hrs, 10 hrs, then 9 hrs daily each period lasting Monday-Thursday of each week, followed by 12 hr daily wear on Fri-Sun
Period: Open Label Dose Optimization
Arm/Group | Group Sequence 1 | Group Sequence 2 | Group Sequence 3 | Group Sequence 4
Started | 6 | 9 | 4 | 7
Completed | 6 | 9 | 4 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Randomized Phase
Arm/Group | Group Sequence 1 | Group Sequence 2 | Group Sequence 3 | Group Sequence 4
Started | 6 | 9 | 4 | 7
Completed | 5 | 8 | 4 | 7
Not Completed | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Sequence 1 | Group Sequence 2 | Group Sequence 3 | Group Sequence 4 | Total
Number analyzed (Participants) | 6 | 9 | 4 | 7 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 9 | 4 | 7 | 26
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 1 | 7
  Male | 4 | 6 | 3 | 6 | 19
Attention Deficit Hyperactivity Disorder (ADHD) Subtype [Number; unit: participants] — There are 3 subtypes of ADHD as defined by the DSM-IV-TR. Inattentive, Hyperactive/Impulsive and combined subtype (hyperactive/impulsive and inattentive). "Other subtype" refers to individuals who are not of the combined subtype but instead are either hyperactive/impulsive or inattentive type.
  participants
    Combined Subtype | 4 | 6 | 3 | 7 | 20
    Other Subtype | 2 | 3 | 1 | 0 | 6
Conner's Global Impression-Parent Scale [Mean (Standard Deviation); unit: scores on scale] — Rating scale filled out by the parents/caregivers. Scale consists of 28 questions divided into four subscales of oppositional problems, cognitive problems, hyperactivity and an ADHD index. Questions scored on a 4 point scale (0-3; 84 points possible), where a higher score indicates more severe symptom presentation.
  scores on scale | 13.7 (7.6) | 20.1 (6.8) | 25 (2.3) | 20.3 (6.7) | 19.78 (6.8)
Attention Deficit Hyperactivity Disorder Rating Scale-IV Total Score [Mean (Standard Deviation); unit: Score on scale] — An 18-item scale corresponding to the 18 items in the DSM-IV-TR that is divided into two subsclaes: hyperactivity/impulsivity and inattentiveness. Items scored on a 4-point frequency scale ranging from 0=never/rarely to 3=very often; 54 points possible with higher score indicating more severe symptoms. Rating scale is filled out by the caregiver.
  Score on scale | 27 (11) | 37 (9.2) | 41 (10.2) | 33.7 (10.6) | 34.7 (11)
Sleep Latency [Mean (Standard Deviation); unit: minutes] — Sleep latency was taken by patient diary which included questions for the caregiver and patient to answer together regarding sleep patterns (time to sleep, duration of sleep, night awakenings, sleep quality)
  minutes | 22.5 (12.6) | 23.3 (21.8) | 54.5 (64.8) | 50.7 (12.4) | 37.8 (27.9)
Total Sleep Time [Mean (Standard Deviation); unit: hours] — Total sleep time was taken by patient diary which included questions for the caregiver and patient to answer together regarding sleep patterns (time to sleep, duration of sleep, night awakenings, sleep quality)
  hours | 9.9 (.9) | 9.5 (.9) | 10.6 (1.2) | 9.6 (1.8) | 9.9 (1.8)
Sleep Quality [Mean (Standard Deviation); unit: Score] — Sleep quality was documented by patient diary which included questions for the caregiver and patient to answer together regarding sleep patterns (time to sleep, duration of sleep, night awakenings, sleep quality). Assessed on a 5 point scale (0-lowest quality; 5-highest quality)
  Score | 4.3 (.8) | 4 (1) | 4 (.8) | 3.1 (.7) | 3.9 (.8)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Latency
Description: Measure by daily subject sleep diary
Time Frame: 9 weeks
Population: All 26 subjects wore the patches for 9, 10, 11 and 12 hour wears. Results are based upon impact of patch wear time on parameter
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- 9 hr Wear: Result for all patients when patch worn for 9 hrs/day
- 10 hr Wear: Result for all patients when patch worn for 10 hrs/day
- 11 hr Wear: Result for all patients when patch worn for 11 hrs/day
- 12 hr Wear: Result for all patients when patch worn for 12 hrs/day
Arm/Group | 9 hr Wear | 10 hr Wear | 11 hr Wear | 12 hr Wear
Number analyzed (Participants) | 26 | 26 | 26 | 26
minutes | 34 [28 to 41] | 34 [27 to 42] | 32 [25 to 35] | 34 [28 to 42]
Statistical Analysis 1: Comparison: 9 hr Wear vs 10 hr Wear vs 11 hr Wear vs 12 hr Wear; Test type: Superiority or Other; p = 0.588, ANOVA; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [0 to 233], Standard Deviation 14

ADVERSE EVENTS:
Arm/Group | Group Sequence 1 | Group Sequence 2 | Group Sequence 3 | Group Sequence 4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 5/9 | 1/4 | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Sequence 1 (N=6) | Group Sequence 2 (N=9) | Group Sequence 3 (N=4) | Group Sequence 4 (N=7)
skin reactions (Skin and subcutaneous tissue disorders) | 2 (4) | 5 (7) | 1 (2) | 4 (6)
Hallucinations (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size, did not permit an examination of more specific differences among patch wear time conditions. Small sample size resulted in weaker randomization to patch wear time sequences that was not completely balanced in baseline covariates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No